CLINICAL TRIAL: NCT03379831
Title: An Observational, Cross-sectional, Multicenter Study Evaluating the Correlation Between Quality of Life and Aerobic Physical Fitness of Patients With a Systemic Right Ventricle.
Brief Title: Correlation Between Quality of Life and Aerobic Physical Fitness of Patients With a Systemic Right Ventricle
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9825
Record Dates: First submitted 2017-11-22; First posted 2017-12-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease
Keywords: systemic right ventricle; quality of life; VO2; oxygen uptake; exercise test; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) is the most common congenital malformations. The right ventricle in the sub-aortic position, or "systemic right ventricle" is one of these complex cardiac diseases. Several studies show that adults with CHD and especially systemic right ventricle have reduced exercise capacity. In addition, studies have shown that there is a correlation between alteration of aerobic physical capacity and alteration of right ventricular systolic function.

Understanding and assessing the determinants of the physical capacity of patients with systemic right ventricles and evaluating their quality of life could allows us to improve their therapeutic management and also to expand patient indications to a program cardiac rehabilitation. This can benefit them on their exercise capacity, their tolerance to exercise and their quality of life.

The aim is to study the correlation between the quality of life and the aerobic physical fitness of patients with a systemic right ventricle and to determine the clinical and paraclinical parameters that have an impact on the aerobic physical fitness of these patients. The quality of life of patients with a systemic right ventricle will be compared to that of the general population.

DETAILED DESCRIPTION:
100 patients will be enrolled in this study. 25 sites will participate to the enrollment, belonging to the French national network for complex congenital heart diseases (M3C) .

Patient is included during his annual medical check-up. Quality of life questionnaire and other examinations are performed during this site visit. Its is a part of his usual care. No supplementary visit, directly related to the research, are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with a right ventricle in the systemic position
* Patient having undergone an annual assessment in accordance with the ESC (European Society of Cardiology) 2010 recommendations: clinical examination, ECG, echocardiography, cardiopulmonary exercise test (with VO2)

Exclusion Criteria:

* Objection of the patient
* Impossibility of performing an exercise test
* Inability to understand and / or complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age, with a right ventricle in the systemic position
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Correlation between the short form SF-36 scores and maximum oxygen uptake (peak VO2) | First day

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Background] Gavotto A, Abassi H, Rola M, Serrand C, Picot MC, Iriart X, Thambo JB, Iserin L, Ladouceur M, Bredy C, Amedro P. Factors associated with exercise capacity in patients with a systemic right ventricle. Int J Cardiol. 2019 Oct 1;292:230-235. doi: 10.1016/j.ijcard.2019.06.030. Epub 2019 Jun 13. PMID 31256996
- [Derived] Padovani P, Werner O, Huguet H, Vaksmann G, Iriart X, Thambo JB, Pierard S, Pasquet A, Domanski O, Godart F, Bredy C, Lefort B, Iserin L, Ladouceur M, Karsenty C, Maragnes P, Moceri P, Cohen S, Hascoet S, Cohen L, Andrianoely M, Combes N, Abassi H, Picot MC, Cornuault L, Amedro P. Health-related quality of life in patients with a systemic right ventricle: the QUALISYSTEMIC study. Eur J Cardiovasc Nurs. 2025 Dec 29;24(8):1260-1271. doi: 10.1093/eurjcn/zvaf156. PMID 40794615